CLINICAL TRIAL: NCT04192474
Title: Clinical Investigation to Evaluate the Performance and Safety of Ambu® aScope™ 4 Cysto and aView™ Urologia for Flexible Cystoscopy
Brief Title: Evaluation of Performance and Safety of Ambu® aScope™ 4 Cysto and aView™ Urologia for Flexible Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ambu A/S (Industry)
Collaborators: QserveCRO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIS-014
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-09

CONDITIONS: Cystoscope; Lower Urinary Tract Symptoms; Bladder Disease
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder Diseases

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, single- arm open-label clinical study on the performance and safety
  * 50% of the patients undergo flexible diagnostic cystoscopy
  * 50% of the patients undergo flexible cystoscopy intervention with endoscopic accessories
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flexible cystoscopy (Other): 50% of the patients undergo flexible diagnostic cystoscopy; 50% of the patients undergo flexible cystoscopy intervention with endoscopic accessories.
  Interventions: Device: Flexible cystoscopy

INTERVENTIONS:
Device: Flexible cystoscopy — Treatment with the investigational device: Ambu® aScope™ 4 Cysto

SUMMARY:
In this study, the new aScope 4 Cysto is used to see if this new single use, flexible cystoscope performs as well as other routinely used flexible cystoscopes. This study will be done in patients who come to the clinic for either a diagnosis of their urethra and bladder or for a small intervention. For an intervention a lesion or tumor is resected, a stent in the ureter is taken out, or an injection in the bladder wall is given. The flexible cystoscope is passed into the urethra and bladder for visual inspection of the bladder and urethra. It will give information on how well the structures of the urinary tract and bladder can be viewed including any abnormalities that are present. If an intervention is performed the aScope 4 Cysto will be used with an endoscopic accessory.

DETAILED DESCRIPTION:
Clinical Phase: pre-CE study

Design: A prospective, multicenter, single- arm open-label clinical study on the performance and safety of Ambu® aScope™ 4 Cysto and aView™ Urologia, a single-use, flexible cystoscope for flexible cystoscopy

Population: Adult subjects (≥ 18 years) undergoing flexible cystoscopy for diagnostic or therapeutic purposes.

Planned Sample Size: A total of 80 patients will result in a maximum (if the true proportion is 50 %) width (i.e. the difference between the point estimate and the upper, or lower, limit of the confidence interval) of the two-sided 95 % confidence interval for the binary variable "Performance level acceptable" to be 11%. This width is considered to be useful in the interpretations of the results from this part of the trial.

Study duration: Screening, procedure and follow-up will take 14 days maximum. A follow-up telephone call at 7 days post procedure is performed to record any adverse events post-procedure.

Planned Trial Period: 3 months

Investigational Device: Ambu® aScope™ 4 Cysto and aView™ Urologia. A pre-CE, single use cystoscope.

ELIGIBILITY:
Inclusion Criteria:

* Adults (males and females), ≥18 years of age or older, presenting for cystoscopy
* Ambulatory with a need to undergo cystoscopy for diagnostic or therapeutic purposes
* Willing to participate in a clinical trial

Exclusion Criteria:

* History of high-grade bladder cancer or carcinoma-in-situ of the bladder, undergoing cystoscopy for follow-up/surveillance purposes
* History of prior bladder/urethral reconstructive surgery
* Presence of symptomatic urinary tract infection (UTI)
* Known unpassable urethral stricture
* Unable to read and/or understand the study requirements
* Unable or unwilling to provide consent to participation in the study
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Performance of the cystoscope | follow up immediately after procedure
  Rate of completion of procedure with Ambu® aScope™ 4 Cysto and aView™ Urologia (yes/no, yes applies to 80% of the procedures)

SECONDARY OUTCOMES:
Overall performance | follow up immediately after procedure
  The overall performance will be further assessed by using a 5-point Likert scale with a minimum of one (=worst possible) to maximum of five (=best possible), to be completed by the investigator that performed the cystoscopy
Procedure time | follow up immediately after procedure
  Procedure time in minutes
Patient Tolerance | follow up immediately after procedure
  Patient tolerance to the procedure measured by 10-points visual analogue scale (VAS) after the flexible cystoscopy. VAS from 0= minimum discomfort and 10=maximum discomfort.
Adverse events | follow up immediately after procedure
  Adverse events evaluation during and immediately after procedure
Adverse events | follow-up at 7 days after procedure
  Adverse events from discharge up to 7 days post-procedure (follow-up call)

CONTACTS AND LOCATIONS:
Locations (2):
- Herlev Hospital, Herlev, Denmark
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No